CLINICAL TRIAL: NCT05435859
Title: Functional Organization of the Superior Temporal Gyrus for Speech Perception
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R01DC012379 (NIH); R01DC012379 (NIH)
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy; Brain Tumor; Speech
MeSH Terms: conditions — Epilepsy; Brain Neoplasms; Speech

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electrocorticography (ECoG) recording during Speech Tasks (Experimental): Participants listened to 25-minute Speech Tasks while ECoG signals for neural activity was recorded during their intraoperative procedure or inpatient hospitalization at the University of California, San Francisco (UCSF).
  Interventions: Behavioral: Speech Tasks

INTERVENTIONS:
Behavioral: Speech Tasks — Listen to 25-minutes of speech sounds in English.

SUMMARY:
The basic mechanisms underlying comprehension of spoken language are still largely unknown. Over the past decade, the study team has gained new insights to how the human brain extracts the most fundamental linguistic elements (consonants and vowels) from a complex and highly variable acoustic signal. However, the next set of questions await pertaining to the sequencing of those auditory elements and how they are integrated with other features, such as, the amplitude envelope of speech. Further investigation of the cortical representation of speech sounds can likely shed light on these fundamental questions. Previous research has implicated the superior temporal cortex in the processing of speech sounds, but little is known about how these sounds are linked together into the perceptual experience of words and continuous speech. The overall goal is to determine how the brain extracts linguistic elements from a complex acoustic speech signal towards better understanding and remediating human language disorders.

DETAILED DESCRIPTION:
Intracranial high-density electrodes make it possible to record neural activity directly from the brain surface with unparalleled spatial and temporal resolution to unravel both local and population encoding of speech sounds. This study proposes to assess speech perception in patients who are undergoing surgery for seizure localization or awake intraoperative brain mapping. Electrode placement is based on the clinical needs of each patient. The research study team will examine the mechanisms of phonetic encoding to reveal both the organization of auditory speech feature selectivity and the distributed population-level processing that give rise to the emergent properties of spoken language perception. The aims of this study seeks to determine the cortical encoding of phonological sequencing (Aim 1), representation of amplitude landmark coding in speech (Aim 2), and the shared and distinct mechanisms for speech and music melody encoding (Aim 3). Together, these aims will advance our understanding of speech encoding in the human brain beyond consonants and vowels, addressing questions pertaining to sequencing, amplitude coding, and auditory specialization. These results should heavily impact current theories of speech processing and, therefore, will have significant implications for understanding and remediating human language disorders.

ELIGIBILITY:
Inclusion Criteria:

* Participants with epilepsy or brain tumors at UCSF undergoing surgical electrode implantation for seizure localization or awake intraoperative brain mapping for resection of brain tumors or epilepsy and
* Participants with electrodes implanted in at least two regions of interest who are willing and able to cooperate with study tasks.

Exclusion Criteria:

* Participants who lack capacity or decline to provide informed consent,
* Participants who have significant cerebral lesions or
* Participants with cognitive deficits that preclude reliable completion of study tasks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Electrocorticography (ECoG) Signals for Neural Activity Identified During Intraoperative Procedure or Inpatient Hospitalization | During Procedure
  Number of participants with ECoG signals for neural activity identified during intraoperative procedure or inpatient hospitalization, between 10-30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Edward F Chang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No